CLINICAL TRIAL: NCT05187026
Title: Electrical Patient Reported Outcome of Prostate Cancer RadioTherapy
Acronym: ePRO-PCaRT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Antti Rannikko, assistant professor, Helsinki University Central Hospital
Other Study IDs: 2067/2016
Record Dates: First submitted 2021-12-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
Keywords: PROM; EPIC-26; electronic; questionnaire; mobile; quality of life; radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EPIC-26 follow-up: All men will receive EPIC-26 in paper and also an electronic version.
  Interventions: Other: electronic PROMs questionnaire

INTERVENTIONS:
Other: electronic PROMs questionnaire — Patients are asked to complete EPIC-26 questionnaire in paper and electronically

SUMMARY:
This is an observational study where prostate cancer related PROMs (EPIC-26) is collected using two different methods (by paper questionnaires and electronically) and patient experience and preference is asked.

DETAILED DESCRIPTION:
Prostate cancer patients that are treated with radiation therapy for local prostate cancer receive EPIC-26 before treatment and during follow-up. EPIC-26 is collected both traditionally using paper questionnaires and electronically. Patients experience and preference for these are asked.

ELIGIBILITY:
Inclusion Criteria:

* cT1-4N0M0, gleason 6-10, PSA < 100, WHO ≤ 2 prostate cancer eligible for radiation therapy
* willing to complete EPIC-26 questionnaires both in paper and electronically
* willing to consent for the study

Exclusion Criteria:

* not able to complete EPIC-26 both in paper and electronically

Ages: 18 Years to 100 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: - local/locally advanced prostate cancer treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-12-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
preference | through study completion, an average of 1 year
  patient preference for type of questionnaire (paper versus electronic)

SECONDARY OUTCOMES:
QoL as measured using the validated EPIC-26 questionnaire | through study completion, an average of 1 year
  Patient QoL after RT (EPIC-26, scale 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Antti S Rannikko, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be shared on the study group website once registered in ClinicalTrials.Gov.
Supporting Information: Study Protocol
Time Frame: Once the study is registered in ClinicalTrials.Gov.
Access Criteria: Publicly available.
URL: http://www.hucc.fi

REFERENCES:
- See also: study group website — http://www.hucc.fi